CLINICAL TRIAL: NCT06426602
Title: Unlocking Functional Communication for Patients With Disorders of Consciousness With Innovative Brain Computer Interface Technology
Brief Title: mindBEAGLE: Unlocking Functional Communication for Patients With Disorders of Consciousness
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Amy Wagner (Other)
Collaborators: The Beckwith Institute (Other)
Responsible Party: Sponsor-Investigator, Amy Wagner, Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY23080022; BECKW/12863 (Other Grant/Funding Number: UPMC Beckwith Institute)
Record Dates: First submitted 2024-01-16; First posted 2024-05-23 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Disorders of Consciousness
Keywords: Coma; Locked-in syndrome; Vegetative state; Unresponsive wakefulness syndrome; Minimally conscious state
MeSH Terms: conditions — Consciousness Disorders; Coma; Locked-In Syndrome; Persistent Vegetative State

STUDY DESIGN:
Intervention Model Description: Single arm Phase 2 experimental device efficacy clinical trial
  To facilitate interpretation of the data generated with this DoC cohort, we will also recruit subjects with locked in syndrome (LIS) receiving care from one or more of our collaborative team and who are not able to communicate via traditional methods but have cognition intact. These patients will follow the same inclusion criteria with the exception of DoC status.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- mindBEAGLE trial participants (Experimental): Patients identified as "disorders of consciousness" admitted to UPMC Rehabilitation Institute will be considered for the trial. As patients will not be able to communicate, health care proxy will provide consent. Participants will undergo 3 trials across 5 days within a 10-day period (2-3 hours each ) to assess if they are responding to the device.
  Interventions: Device: mindBEAGLE daily device use

INTERVENTIONS:
Device: mindBEAGLE daily device use — If participants are considered responsive, they will continue to use the device daily for the remainder of their stay at inpatient rehab, or until they regain consciousness.

SUMMARY:
The goal of this clinical trial is to test how effective the mindBEAGLE device is in allowing people who are unconscious (due to a brain injury or other condition) to communicate using brain waves to answer Yes/No questions. Participants will wear a cap that will be connected to a computer that measures brain waves, wrist bands that vibrate at different strengths, and ear phones that create different levels of loud tones and will be asked to associate Yes/No answers with the vibrations or tones. They will also be asked to "think about" moving different parts of their body to answer Yes or No. The mindBEAGLE device has already been proven effective for this kind of communication in a previous study, and the study team would like to trial it on a population of unconscious people who enter the UPMC Rehabilitation Institute to see if patients are able to be trained to use the device as part of their everyday inpatient rehabilitation until they are discharged, or until they are able to regain consciousness.

DETAILED DESCRIPTION:
The team's research reflects an integrated clinical and research team who will characterize and implement an aggressive and innovative approach using brain-computer interface (BCI) technology for Disorders of Consciousness (DoC) evaluation, prognostication, and rehabilitation care. The work proposed strives for equity in accessing healthcare systems and technology effectively, even among vulnerable individuals with profound levels of disability due to their DoC state.

The "gold-standard" for assessing cognitive capacity among patients with DoC relies on behavioral response observations and neuroimaging modalities. However, these approaches underestimate patients' capabilities. The current problem is that without other clinical data, rehabilitation teams rely solely on observable behavioral changes in patients' awareness of their environment in order to treat and improve communication. The project's challenge rests with implementing BCI focused assistive technology that identifies a unique and specific electrophysiological biomarker of cognitive and communication capacities that cannot be tapped using current clinical tools. If successful, this approach will allow clinical teams to initiate treatment and communication, avoiding therapeutic delays arising from traditional methods that require behavioral indicators needed to participate in functional communication.

The P300 wave is a positive deflection in the human event-related potential. It is most commonly elicited in an "oddball" paradigm when a subject detects an occasional "target" stimulus in a regular train of standard stimuli.

This project will compare standard awareness training methods used at the UPMC RI Brain Injury program with novel BCI research by using mindBEAGLE, a suite of P300 paradigms (vibrations, sound tones, and mental visualization) used for cognitive and communication assessment and treatment. European studies using the mindBEAGLE system with DoC patients reveal patients' cognitive and communication capabilities that impact current functional assessment and influence prognostication and recovery. The mindBEAGLE gives additional diagnostic data to enhance clinical neuroscience practice by showing reactions to stimuli that benefit from electroencephalogram (EEG) P300 use. However, clinical neuroscience implementation studies have not been conducted. Armed with more detailed and accurate assessments from this study, the investigators are confident that the clinical teams will be able to offer exciting rehabilitation treatments designed by UPMC RI treatment teams, patients, and families that leverage the mindBEAGLE interface for functional communication. Specifically, the EEG-based mindBEAGLE BCI suite will provide a practical platform for cognitive assessment of command following and a communication system for patients with DoC that will allow the research teams to offer more intensive, multidimensional rehabilitation treatments that meet the UPMC ideal of Life Changing Medicine.

ELIGIBILITY:
Inclusion Criteria:

* Age 16-65
* Medically able to tolerate Disorders of Consciousness (DoC) rehabilitation program as determined by UPMC Physicians
* Locked in Syndrome (LIS) patients who show clinical evidence of intact cognition via some form of alternative communication methods
* Clinically assessed capacity for functional improvement in the rehabilitation environment
* Measuring improvements with pharmacological stimulation (using JFK Coma Recovery Scale)
* Electrophysiological prognostic testing confirming brain activity.

Exclusion Criteria:

* Coma
* Bilateral non-response with standard electrophysiological studies
* Medical instability
* Open scalp wound

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Neural and Multisensory DOC mindBEAGLE Initial Classification Accuracy Assessment | 18 months
  The ability to answer Yes/No questions at over above 40% accuracy using 1 of the following paradigms:
  1. auditory evoked potentials;
  2. vibro-tactile stimulation with 2 tactors;
  3. vibro-tactile stimulation with 3 tactors;
  4. vibro-tactile stimulation with 7 tactors;
  5. motor imagery.
DOC mindBEAGLE Communication Assessment | 18 months
  Among DOC patients who pass initial classification assessment: ability to communicate yes/no questions at or above 40% accuracy with one of the two P300 paradigms.
  mindBEAGLE P300 paradigm #1
  1. Baseline - No response to yes/no questions
  2. Change in baseline - Response to yes/no questions using mindBEAGLE
  mindBEAGLE P300 paradigm #2
  1. Baseline - 0% accuracy on yes/no questions
  2. Change in baseline - 60% or higher in response to yes/no questions.
Acceptability of mindBEAGLE treatment by clinical staff. | Within 2 weeks Post-intervention
  Clinicians agree that mindBEAGLE is feasible to implement with DOC patients in the inpatient setting.
Acceptability of mindBEAGLE treatment by families of DOC patients. | Within 2 weeks Post-intervention
  Family/Caregivers of DOC patient agree that the mindBEAGLE was beneficial.

CONTACTS AND LOCATIONS:
Overall Officials: Amy Wagner, M.D., Principal Investigator — University of Pittsburgh; Katherine Hill, Ph.D., Principal Investigator — University of Pittsburgh
Locations (2):
- United States (2):
  - UPMC Center for Assistive Technology, Pittsburgh, Pennsylvania
  - UPMC Rehabilitation Institute, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
It is possible that the investigators may use the information obtained from this study in other future research studies. All information disseminated to outside collaborators or entities will be done in a de-identified manner so as to mitigate a breach of confidentiality and protect PHI/PII. Data will be coded using unique identifying numbers that do not contain PII. Any links to PII will be kept locally but will not be disseminated to outside collaborators.
  Any data shared with outside institutions or collaborators will be conducted under the guidelines of an approved data use agreement between the University of Pittsburgh and the collaborating entity. This includes any plans to publish published peer-reviewed manuscripts.

REFERENCES:
- [Background] Kondziella D, Amiri M, Othman MH, Beghi E, Bodien YG, Citerio G, Giacino JT, Mayer SA, Lawson TN, Menon DK, Rass V, Sharshar T, Stevens RD, Tinti L, Vespa P, McNett M, Venkatasubba Rao CP, Helbok R; Curing Coma Campaign Collaborators. Incidence and prevalence of coma in the UK and the USA. Brain Commun. 2022 Sep 1;4(5):fcac188. doi: 10.1093/braincomms/fcac188. eCollection 2022. PMID 36132425
- [Background] Godbolt AK, Deboussard CN, Stenberg M, Lindgren M, Ulfarsson T, Borg J. Disorders of consciousness after severe traumatic brain injury: a Swedish-Icelandic study of incidence, outcomes and implications for optimizing care pathways. J Rehabil Med. 2013 Sep;45(8):741-8. doi: 10.2340/16501977-1167. PMID 24002309
- [Background] van der Wal D. Codependency: a concomitant field of interest in research into the phenomenon caring. Curationis. 1996 Dec;19(4):40-2. doi: 10.4102/curationis.v19i4.1335. PMID 9283342
- [Background] Torres-Saavedra PA, Winter KA. An Overview of Phase 2 Clinical Trial Designs. Int J Radiat Oncol Biol Phys. 2022 Jan 1;112(1):22-29. doi: 10.1016/j.ijrobp.2021.07.1700. Epub 2021 Aug 4. PMID 34363901